CLINICAL TRIAL: NCT07026136
Title: Application of Blended Learning Model to Improve the Communication Skills of Nursing Students and New Nurses With the Elderly: Development and Effectiveness Verification
Brief Title: Blended Learning to Enhance Elderly Communication Skills in Nursing Students and New Nurses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CMUH111-REC1-110
Record Dates: First submitted 2025-04-29; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Communication; Elderly Patients
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: Hybrid method course of learning effective communicating skill
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid Learning: Digital Modules + AI Chatbot Support (Experimental): Participants in this arm will complete a 60-minute hybrid learning session using online digital textbooks developed by the research team. Content includes modules on aging knowledge, empathy techniques, communication barriers, and simulated scenario-based dialogues. Each module is followed by an online quiz. After the session, learners can continue practicing with an AI chatbot that provides personalized guidance and simulated dialogue practice.
  Interventions: Other: Hybrid Digital Learning with AI Chatbot for Geriatric Communication
- Traditional Learning: Printed Educational Materials (Active Comparator): Participants in this arm will study the same instructional content using printed materials within a 60-minute session. The content parallels that of the digital modules but is provided in static written format, without multimedia or chatbot interaction.
  Interventions: Other: Traditional Learning: Printed Educational Materials

INTERVENTIONS:
Other: Hybrid Digital Learning with AI Chatbot for Geriatric Communication — A web-based, self-directed learning program integrated with a conversational AI chatbot. The chatbot reinforces learning and allows for flexible post-training practice.
  Arms: Hybrid Learning: Digital Modules + AI Chatbot Support
Other: Traditional Learning: Printed Educational Materials — Traditional teaching materials, printed document including structured readings on aging knowledge, empathy, communication barriers, and case-based communication strategies with older adults.
  Arms: Traditional Learning: Printed Educational Materials

SUMMARY:
The study will recruit new nurses from the hospital to evaluate the effectiveness of learning communicating skills in elderly care through a hybrid learning model. Participants will be randomly assigned to either an experimental group receiving hybrid method course or a control group using written materials, with both groups participating in a 60-minute educational session. The research will employ a multi-stage assessment approach, beginning with a pre-test to measure baseline knowledge of aging, attitudes toward older adults, willingness to serve the elderly, and communication skills. Immediately following the intervention, participants will complete a post-test, with a follow-up delayed assessment conducted three months later to evaluate knowledge retention. Clinical preceptors will systematically assess the nurses' elderly communication skills using a standardized rating scale. To gain deeper insights, selected nurses will also participate in qualitative interviews, sharing their learning experiences, reflections, and recommendations for improving the teaching materials, thereby providing a comprehensive understanding of the training's effectiveness and potential areas of enhancement.

DETAILED DESCRIPTION:
This study is a randomized controlled trial designed to evaluate the effectiveness of a hybrid learning model communication training program for newly recruited nurses interacting with older adults. The intervention group receives a self-directed learning experience using an online multimedia module and an AI chatbot learning assistant, while the control group studies equivalent content through printed educational materials. The training aims to enhance nurses' knowledge of aging, improve attitudes toward older adults, increase willingness to serve the elderly, and develop geriatric communication skills.

The digital course content includes five core themes: (1) knowledge related to aging, (2) application of empathy, (3) the impact of hospitalization on older adults and communication barriers, (4) fundamental principles of elderly communication, and (5) simulated scenario-based dialogues. Each unit is under 10 minutes and followed by an online quiz. Participants may continue practicing using an AI chatbot tutor that reinforces learning.

Participants are randomly assigned in a 1:1 ratio stratified by gender and educational background. Following baseline assessments, the intervention is conducted during the fourth day of an onboarding training program. The post-test is planned to be done immediately after the 60-minute learning session, and follow-up assessments are conducted one, two, and three months later to evaluate knowledge retention and real-world skill application. Quantitative outcome measures include pre-post changes in: knowledge of aging questionnaire, attitudes toward older adults questionnaire, willingness to care for elderly questionnaire, self-reported and preceptor-assessed geriatric communication skills questionnaire, motivation for learning via instructional material.

In addition to self-report questionnaires, trained clinical preceptors assess geriatric communication skills during actual clinical settings using the KEECC Checklist (Kalamazoo Essential Elements Communication Checklist).

A final qualitative component includes semi-structured interviews with 10 participants from the experimental group, selected until data saturation is reached, to explore learning experiences and gather feedback on the instructional design.

This mixed-method study aims to provide evidence for scalable, technology-enhanced training solutions that prepare early-career nurses for competent and compassionate elder care communication.

ELIGIBILITY:
Inclusion Criteria:

* At least 20 years old
* Graduated from a nursing school
* Full-time employee
* Less than six months of nursing work experience
* Working in a medical ward

Exclusion Criteria:

* Job nature does not involve direct patient contact, such as working in the supply room.
* Not engaged in clinical nursing work, such as a research assistant.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Knowledge of Aging Questionnaire Score | Baseline (Pre-test): Prior to intervention. Immediate Post-test: Directly after the 60-minute learning session. First Follow-up: 1 month after intervention. Second Follow-up: 2 months after intervention. Third Follow-up: 3 months after intervention.
  * Instrument: 19-item scale developed by Hsieh & Yang (2009)
  * Score range: 19-95 (Likert 5-point scale)
  * Higher scores indicate: Greater knowledge of aging (biological, psychological, and social aspects)
Change in Kogan's Attitudes Toward Older People (KAOP) Scale Score | Baseline (Pre-test): Prior to intervention. Immediate Post-test: Directly after the 60-minute learning session. First Follow-up: 1 month after intervention. Second Follow-up: 2 months after intervention. Third Follow-up: 3 months after intervention.
  * Instrument: 34-item Chinese version by Yeh et al., 2018
  * Score range: 34-204 (Likert 6-point scale, with reverse-coded items)
  * Higher scores indicate: More positive attitudes toward older adults
Change in Willingness to Serve Older Adults Scale Score | Baseline (Pre-test): Prior to intervention. Immediate Post-test: Directly after the 60-minute learning session. First Follow-up: 1 month after intervention. Second Follow-up: 2 months after intervention. Third Follow-up: 3 months after intervention.
  * Instrument: 16-item scale by Hsieh & Yang (2009)
  * Score range: 16-80(Likert 5-point scale)
  * Higher scores indicate: Greater willingness to provide care or service to older adults
Change in Self-Reported Communication Skills Scale Score | Baseline (Pre-test): Prior to intervention. Immediate Post-test: Directly after the 60-minute learning session. First Follow-up: 1 month after intervention. Second Follow-up: 2 months after intervention. Third Follow-up: 3 months after intervention.
  * Instrument: Adapted from Canary & Spitzberg's CAE, modified by Chen (2017)
  * Score range: 28-168 (Likert 6-point scale)
  * Higher scores indicate: Higher perceived appropriateness and effectiveness in communication
Change in Kalamazoo Essential Elements Communication Checklist (KEECC) Score | Baseline (Pre-test): Prior to intervention. Immediate Post-test: Directly after the 60-minute learning session. First Follow-up: 1 month after intervention. Second Follow-up: 2 months after intervention. Third Follow-up: 3 months after intervention.
  * Instrument: 7-domain, 5-point checklist adapted for elder-care scenarios
  * Score range: 7-35
  * Rated by: Clinical preceptors after observed interactions
  * Higher scores indicate: Better objective communication performance

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Tzeng, Taichung
  - Ya-Ling Tzeng, Taichung